CLINICAL TRIAL: NCT06676007
Title: A Multicenter Open Label Prospective Study on Early Initiation of Targeted-release Formulation of Budesonide in Patients With Primary IgA Nephropathy
Brief Title: A Multi-center Open Label Prospective Study on Early Initiation of Targeted-release Formulation of Budesonide in Patients With Primary IgA Nephropathy
Status: Recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Guisen Li, Director of Nephrology Department, Sichuan Provincial People's Hospital
Other Study IDs: NEF-EM-004
Record Dates: First submitted 2024-10-31; First posted 2024-11-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: IgA Nephropathy (IgAN); Early Initial Therapy
Keywords: IgA Nephropathy (IgAN); Nefecon; multi-center; Early Initial Therapy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — UPCR, eGFR, blood chemistry, blood routine, urine routine, 24-hour Urine Protein Quantitation, etc..
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gd-IgA1 test — collect and test Gd-IgA1 test in enrolled subjects

SUMMARY:
To observe of the efficacy and safety of early initiation of budesonide enteric coated capsules in the treatment of primary IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Target patients aged 18-75, including those aged 18 and 75
2. Primary IgA nephropathy diagnosed by renal biopsy within 3 months
3. eGFR≥30ml/min/1.73m2
4. 24-hour urine protein ≥ 1.0g/d, or UPCR ≥ 0.8 g/g
5. Sign informed consent

Exclusion Criteria:

1. Including but not limited to secondary IgAN caused by allergic purpura, systemic lupus erythematosus, cirrhosis, rheumatoid arthritis, and ankylosing spondylitis
2. Patients who have received kidney transplantation or dialysis
3. Patients with other glomerular diseases (such as C3 glomerular disease and/or diabetes nephropathy) and nephrotic syndrome (i.e. proteinuria>3.5 g/d, serum albumin<3.0 g/dl, with or without edema)
4. Patients with acute, chronic, or potential infectious diseases, including hepatitis, tuberculosis, human immunodeficiency virus, and chronic urinary tract infections
5. Patients with type 1 or type 2 diabetes diagnosed and poorly controlled (HbA1c>8%)
6. Patients with a history of unstable angina, grade III or IV congestive heart failure, and/or clinically significant arrhythmias
7. Patients with poor blood pressure control (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90mmHg)
8. Patients diagnosed with malignant tumors within the past 5 years
9. Patients with known glaucoma, known cataracts, and/or a history of cataract surgery
10. Gastrointestinal diseases that may interfere with the study of drug efficacy or release, such as peptic ulcer disease, inflammatory bowel disease, and chronic diarrhea
11. Patients with severe adverse reactions to steroids in the past, including psychiatric symptoms
12. Patients who have received systemic immunosuppressive drug treatment within 3 months prior to enrollment
13. Patients who have received any systemic GCS treatment within the past 3 months prior to enrollment
14. Patients taking potent cytochrome P450 3A4 inhibitors (CYP3A4)
15. Current or previous (within the past 2 years) alcoholism or drug abuse;
16. Expected lifespan<5 years
17. During the study treatment period and 3-month follow-up period, women who are pregnant, breastfeeding, or unwilling to use highly effective contraception (contraception is only required for women with fertility potential)
18. Researchers believe that patients who are not suitable for treatment with Nefecon

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female, aged 18 to 75 years, diagnosed with primary IgA nephropathy through renal biopsy within 3 months, with eGFR ≥ 30ml/min/1.73m2, 24-hour urinary protein ≥ 1.0g/d, and blood pressure<140/90mmHg
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The changes in proteinuria levels | about 12 months
  To evaluate the changes in proteinuria levels of the target patient in the 12th month compared to baseline
Number of Participants With clinical significant Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment. | about 12 months
  Safety event

SECONDARY OUTCOMES:
Evaluate the changes in eGFR of target patients at the 12th month compared to baseline | about 12 months
Evaluate the changes in microscopic hematuria of the target patient at the 12th month compared to baseline | about 12 months
Assess the incidence of composite renal endpoint events (eGFR decreased by 40% from baseline or ESKD) in target patients | about 12 months
Assess the incidence of ESKD (eGFR<15ml/min/1.73m2) in target patients at the 12th month | about 12 months
Evaluate the proportion of target patients with a 40% decrease in eGFR compared to baseline at the 12th month | about 12 months
Evaluate the proportion of target patients whose average urinary protein level decreased by 50% from baseline in the 12th month | about 12 months
Evaluate the changes in serum and urine proteomics and metabolomics of the target patient in the 12th month | about 12 months

OTHER OUTCOMES:
Evaluate the changes in GD-IgA1 levels of the target patient at 12 months compared to baseline. | about 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No